CLINICAL TRIAL: NCT03064997
Title: Assessment of the Impact of Prebiotic Synergy 1 on the Intestine Permeability, Clinical Symptoms, and Selected Biochemical and Nutritional Parameters in the Children With Celiac Disease on a Gluten-free Diet
Brief Title: Prebiotic as a Supplement of Gluten-free Diet in the Management of Celiac Disease in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polish Academy of Sciences (Other)
Collaborators: University of Warmia and Mazury (Other)
Responsible Party: Principal Investigator, Urszula Krupa-Kozak, Ph.D., Polish Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IAR&FR internal project 20
Record Dates: First submitted 2017-02-16; First posted 2017-02-27 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Celiac Disease
Keywords: prebiotic; pediatric patients; health status; intestine permeability
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic Synergy 1-supplemented GFD (Active Comparator): The application of a prebiotic Synergy 1 together with a strict gluten-free diet
  Interventions: Dietary Supplement: Synergy 1
- Placebo-supplemented GFD (Placebo Comparator): The application of a placebo together with a strict gluten-free diet
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synergy 1 — a daily dose: 7 g/day of Synergy1 (oligofructose enriched inulin) consumed for 12 weeks together with a strict gluten-free diet
  Arms: Prebiotic Synergy 1-supplemented GFD
Dietary Supplement: Placebo — a daily dose: 7 g/day of placebo (maltodextrin) consumed for 12 weeks together with a strict gluten-free diet
  Arms: Placebo-supplemented GFD

SUMMARY:
Prebiotics are known as substances affecting beneficially the organism by restoring the intestinal microbiota balance, stabilizing the intestinal barrier and modulating the endocrine and immune functions. In many persons suffering from celiac disease (CD), despite a gluten-free diet (GFD), an impaired intestinal barrier functionality, accompanied by altered intestinal microbiota and ongoing intestinal inflammation is observed. For these reasons, prebiotic could be a promising and low-risk adjuvant in the dietetic management of CD. It was hypothesize that prebiotic preparation Synergy 1 consumed by CD children as a supplement of a GFD will affect beneficial the intestinal permeability and intestinal microbiota without side effects.

DETAILED DESCRIPTION:
Prebiotics, including inulin-type fructans (ITFs) are a group of the naturally occurring plant carbohydrates stored in various amounts in tubers, bulbs and tuberous roots of several edible fruits and vegetables and in particularly large amounts in the tubers of Helianthus tuberosus (Jerusalem artichoke) and Cichorium intybus (chicory). Because of their unique structural properties, they are not hydrolyzed by the enzymes of the upper intestinal digestive tract and reach the colon unchanged, therefore are classified as prebiotics. Prebiotics are defined as selectively fermented ingredients that allow specific changes in the composition and/or balance of the microbiota. ITFs, particularly the mixture of short- and long-chain polymers, indicate several beneficial effects, including the positive changes in the histological picture of the intestine (proliferation in the crypts and Goblet cells, longer intestinal villi) and modulation of the endocrine and immune functions. Moreover, they have a great potential as agents improving or maintaining a balanced intestinal microbiota both in the lumen and at the mucosal surface, to one in which bifidobacteria and lactobacilli come to greater prominence. This, so-called healthier flora, should provide increased resistance to gut infections and may also have immuno-modulatory properties. Until now, inulin and fructooligosaccharide (FOS) have been tested mainly in animal models of inflammatory bowel diseases (IBD). Reports on animal colitis model suggests that prebiotics have the anti-inflammatory properties as they reduce the inflammation symptoms, along with the increase in bifidobacteria or lactobacilli number, and in some reports, the increase in the concentration of butyrate in the gut.

Prebiotics are known as substances affecting beneficially the organism by restoring the intestinal microbiota balance, stabilizing the intestinal barrier and modulating the endocrine and immune functions. In many persons suffering from celiac disease (CD), despite a gluten-free diet (GFD), an impaired intestinal barrier functionality, accompanied by altered intestinal microbiota and ongoing intestinal inflammation is observed. For these reasons, prebiotics could be a promising and low-risk adjuvant in the dietetic management of CD. It was hypothesized that Synergy 1 consumed by CD children as a supplement of a GFD will affect beneficial the intestinal permeability and intestinal microbiota without side effects. The primary objective of this randomized placebo-controlled study was to determine the effect of 3-months consumption of Synergy 1 versus placebo, as the supplements of a GFD, on the intestinal permeability in CD children, in particular on the concentration of the intestinal fatty acid binding protein (iFABP) as a biomarker of intestinal permeability. The secondary objective was to determine the effect of Synergy 1 versus placebo applied in GFD on the changes in the gut microbiota quantity and metabolism in CD children.

ELIGIBILITY:
Inclusion Criteria:

* celiac disease
* treatment with gluten-free diet for at least 6 months
* general good health
* the written informed consent to participate the study

Exclusion Criteria:

* participation in another study involving prebiotic and/or probiotic preparations, or intention to use such products during the course of the study
* other gastrointestinal diseases
* received antibiotics in the previous month
* use of dietary supplements containing prebiotic or/and probiotic within the previous month
* bad or average overall health

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the intestinal permeability | 6 months
  Changes in the concentration of intestinal fatty acid binding protein (iFABP) as a biomarker of intestinal permeability will be determined

SECONDARY OUTCOMES:
Assessment of the advers events | 6 months
  A number of participants with adverse events related to the treatment will be recorded
Analysis of the concentration of the short chain fatty acids (SCFAs) | 6 month
  Changes in the concentration and a profile of the short chain fatty acids (SCFAs) using gas chromatography
Molecular characteristic of faecal microbiota | 6 month
  Quantitative characteristics of faecal bacteria will be conducted with the real-time polymerase chain reaction (RT-PCR) technique and group-specific primers. Population level of Bifidobacterium, Bacteroides, Clostridium coccoides, C. leptum and E. coli groups will be determined among others.

CONTACTS AND LOCATIONS:
Overall Officials: Urszula Krupa-Kozak, Ph.D, Principal Investigator — Institute of Animal Reproduction and Food Reseach, Polish Academy of Sciences in Olsztyn; Elżbieta Jarocka-Cyrta, MD, Ph.D, Principal Investigator — Department of Clinical Pediatrics, Faculty of Medical Sciences, University of Warmia and Mazury
Locations (2):
- Poland (2):
  - Regional Specialized Children'S Hospital, Olsztyn
  - Institute of Animal Reproduction and Food Research, Polish Academy of Sciences in Olsztyn, Olsztyn

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drabinska N, Jarocka-Cyrta E, Ratcliffe NM, Krupa-Kozak U. The Profile of Urinary Headspace Volatile Organic Compounds After 12-Week Intake of Oligofructose-Enriched Inulin by Children and Adolescents with Celiac Disease on a Gluten-Free Diet: Results of a Pilot, Randomized, Placebo-Controlled Clinical Trial. Molecules. 2019 Apr 5;24(7):1341. doi: 10.3390/molecules24071341. PMID 30959740
- [Result] Drabinska N, Jarocka-Cyrta E, Zlotkowska D, Abramowicz P, Krupa-Kozak U. Daily oligofructose-enriched inulin intake impacts bone turnover markers but not the cytokine profile in pediatric patients with celiac disease on a gluten-free diet: Results of a randomised, placebo-controlled pilot study. Bone. 2019 May;122:184-192. doi: 10.1016/j.bone.2019.03.001. Epub 2019 Mar 3. PMID 30840918
- [Result] Ferus K, Drabinska N, Krupa-Kozak U, Jarocka-Cyrta E. A Randomized, Placebo-Controlled, Pilot Clinical Trial to Evaluate the Effect of Supplementation with Prebiotic Synergy 1 on Iron Homeostasis in Children and Adolescents with Celiac Disease Treated with a Gluten-Free Diet. Nutrients. 2018 Nov 21;10(11):1818. doi: 10.3390/nu10111818. PMID 30469412
- [Result] Drabinska N, Krupa-Kozak U, Abramowicz P, Jarocka-Cyrta E. Beneficial Effect of Oligofructose-Enriched Inulin on Vitamin D and E Status in Children with Celiac Disease on a Long-Term Gluten-Free Diet: A Preliminary Randomized, Placebo-Controlled Nutritional Intervention Study. Nutrients. 2018 Nov 15;10(11):1768. doi: 10.3390/nu10111768. PMID 30445682
- [Result] Drabinska N, Krupa-Kozak U, Ciska E, Jarocka-Cyrta E. Plasma profile and urine excretion of amino acids in children with celiac disease on gluten-free diet after oligofructose-enriched inulin intervention: results of a randomised placebo-controlled pilot study. Amino Acids. 2018 Oct;50(10):1451-1460. doi: 10.1007/s00726-018-2622-7. Epub 2018 Jul 24. PMID 30043079
- [Result] Drabinska N, Jarocka-Cyrta E, Markiewicz LH, Krupa-Kozak U. The Effect of Oligofructose-Enriched Inulin on Faecal Bacterial Counts and Microbiota-Associated Characteristics in Celiac Disease Children Following a Gluten-Free Diet: Results of a Randomized, Placebo-Controlled Trial. Nutrients. 2018 Feb 12;10(2):201. doi: 10.3390/nu10020201. PMID 29439526
- [Derived] Krupa-Kozak U, Drabinska N, Jarocka-Cyrta E. The effect of oligofructose-enriched inulin supplementation on gut microbiota, nutritional status and gastrointestinal symptoms in paediatric coeliac disease patients on a gluten-free diet: study protocol for a pilot randomized controlled trial. Nutr J. 2017 Aug 22;16(1):47. doi: 10.1186/s12937-017-0268-z. PMID 28830428